CLINICAL TRIAL: NCT01320072
Title: Diagnosis of Aspirin Hypersensitivity in Aspirin Exacerbated Respiratory Disease Using a Safe, Low Dose Aspirin Challenge
Brief Title: Diagnosis of Aspirin Hypersensitivity in Aspirin Exacerbated Respiratory Disease
Acronym: ASAS
Status: Terminated | Type: Observational
Why Stopped: Study discontinued and closed out by IRB. PI left the institution.
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 10-01-002
Record Dates: First submitted 2011-03-17; First posted 2011-03-22 (Estimated); Results first posted 2016-04-05 (Estimated); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Asthma, Aspirin-induced
Keywords: aspirin; asthma; diagnosis; prostaglandins; leukotrienes
MeSH Terms: conditions — Asthma, Aspirin-Induced; Asthma; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine, peripheral blood mononuclear cells, plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Aspirin-sensitive asthmatics: asthma patients with aspirin allergy
- aspirin-tolerant asthmatics: asthma patients without aspirin allergy

SUMMARY:
To diagnose aspirin hypersensitivity in asthmatics by using and safe, low-dose aspirin oral challenge.

Hypothesis 1: A low dose of oral ASA (20 or 40 mg) will induce significantly different concentrations of arachidonic acid metabolites in ASA-sensitive asthmatics as compared to ASA-tolerant asthmatics.

Hypothesis 2: The low dose (20 or 40 mg) ASA challenge will be well tolerated by ASA-sensitive asthmatics.

DETAILED DESCRIPTION:
This research study is being conducted within the established Airway Research Group at Montefiore Medical Center and Albert Einstein College of Medicine in Bronx, NY. The patient population in the Bronx has one of the highest asthma prevalences in the country. Thus, our study participants are being recruited among the population most in need of a better understanding of the disease process.

Visits 1 and 2: Low-dose challenge with 20 mg and 40 mg of ASA. ASA will be administered orally to participants in both groups: 20 mg at Visit 1 and 40 mg at Visit 2. Visits will take place at least 1 week apart. Blood and urine will be collected at several time points.

Visit 3: Oral graded ASA challenge will be performed to confirm or rule out the presence of ASA-hypersensitivity. This visit will take place at least 1 week after Visit 2. Both groups will undergo an oral graded ASA challenge as per earlier described protocol. Urine and plasma will be collected from the patients at several time points. Hypersensitivity reactions will be defined in four different ways: a) decline in forced expiratory volume in 1 second (FEV1) of at least 15% combined and naso-ocular reaction; b) 20% decline in FEV1; c) isolated naso-ocular reactions; d) isolated cutaneous reactions (hives and swelling). Patients with reactions will be treated according to their symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Participants of both sexes aged 18 years and older.
2. Patients with a history of ASA-induced asthma who had at least one asthma attack after ingestion of aspirin or other NSAIDs.
3. Patients with a history of ASA-tolerant asthma who had been occasionally using aspirin or other NSAIDs without any adverse reactions.

Exclusion Criteria:

1. Mental or legal incapacitation, or significant emotional problems, or a history of psychiatric disorders at the time of the enrollment.
2. Pregnancy or breastfeeding at the time of enrollment.
3. History of a severe anaphylactic reaction precipitated by ASA and/or other NSAIDs (such as ibuprofen, naproxen, indomethacin, Advil, Aleve, Motrin, diclofenac, etc.).
4. History of a severe bronchospasm precipitated by ASA and/or other NSAIDs requiring an endotracheal intubation.
5. Chronic kidney disease (a calculated GFR based on the Modification of Diet in Renal Disease (MDRD) equation is < 60 mL/min/1.73 sq.meter).
6. Chronic liver disease by history and/or abnormal liver function tests (SGOT and SGPT ≥ 3 times above upper normal range).
7. Baseline FEV1 < 70% (or < 1.5 L) of predicted, or an exacerbation of asthma in the 6 weeks preceding the study.
8. An active infectious disease.
9. Anemia that requires work-up, black stools, active bleeding.
10. A history of gastrointestinal bleeding due to aspirin or other NSAIDS, gastritis, or duodenal ulcer not proven to be due to Helicobacter pylori.
11. A history of hemophilia or any other bleeding disorder.
12. Unstable angina.
13. Participants taking aspirin and or other NSAIDs at the time of the study visits.
14. Participants taking leukotriene receptors inhibitors or 5-lypooxygenase (5-LO) inhibitors at the time of the study visits.
15. In addition, participants taking one or more of the following drugs intake last 14 days prior to the enrollment will be excluded: lithium, warfarine, enoxaparin, heparin, dalteparin, fluconazole, ketotifen. Short-acting antihistamines should be stopped 5 days before the challenge; long-acting antihistamines should be stopped 1 week prior to the challenge.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Allergy/Immunology clinic population in Bronx, NY
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2022-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elina Jerschow, MD, Principal Investigator — Attending physician
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
no, patients signed informed consent that allowed us to collect data for the present study but not to share the data

REFERENCES:
- [Background] Jerschow E, Ren Z, Hudes G, Sanak M, Morales E, Schuster V, Spivack SD, Rosenstreich D. Utility of low-dose oral aspirin challenges for diagnosis of aspirin-exacerbated respiratory disease. Ann Allergy Asthma Immunol. 2016 Apr;116(4):321-328.e1. doi: 10.1016/j.anai.2015.12.026. Epub 2016 Jan 25. PMID 26822279

RESULTS

PARTICIPANT FLOW:
Groups:
- Aspirin-sensitive Asthmatics: Patients with aspirin exacerbated respiratory disease, N=16
- Aspirin-tolerant Asthmatics: Aspirin tolerant asthma patients, N=13
Period: Overall Study
Arm/Group | Aspirin-sensitive Asthmatics | Aspirin-tolerant Asthmatics
Started | 16 | 13
Completed | 16 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Aspirin-sensitive Asthmatics: patients with aspirin exacerbated respiratory disease
- Aspirin-tolerant Asthmatics: aspirin-tolerant patients with asthma
- Total: Total of all reporting groups
Arm/Group | Aspirin-sensitive Asthmatics | Aspirin-tolerant Asthmatics | Total
Number analyzed (Participants) | 16 | 13 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 13 | 29
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (3.2) | 42.6 (2.4) | 40.3 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 8 | 17
  White | 7 | 4 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 13 | 29

OUTCOME MEASURES:

1. Primary Outcome: Eicosanoid Metabolites Concentration
Description: eicosanoid metabolites concentration in plasma and urine 2 h post ASA challenge
Time Frame: 2 hours
Measure: Mean (Standard Error); unit: log-pg/mg creatinine
Arm/Group | Aspirin-sensitive Asthmatics | Aspirin-tolerant Asthmatics
Number analyzed (Participants) | 16 | 13
log-pg/mg creatinine | 6.91 (0.15) | 5.8 (0.12)

2. Secondary Outcome: Treatment-Related Adverse Events
Description: Adverse reactions defined as bronchospasm requiring endotracheal intubation. The adverse reactions will be assessed through a post challenge follow-up with the patient at baseline and 24 hours after the challenge
Time Frame: 24 hours after the challenge
Measure: Number; unit: participants
Arm/Group | Aspirin-sensitive Asthmatics | Aspirin-tolerant Asthmatics
Number analyzed (Participants) | 16 | 13
participants | 0 | 0

3. Secondary Outcome: Change in Forced Expiratory Volume in One Second (FEV1) in Aspirin Exacerbated Respiratory Disease (AERD) Patients
Description: We will assess FEV1% change from baseline at 12 months in AERD patients who have been on aspirin treatment for 12 months (current standard of care)
Time Frame: 12 months
Population: AERD patients will continue aspirin treatment for 12 months and the change from baseline in their FEV1% predicted will be monitored during this time
Measure: Mean (Standard Error); unit: change in percent predicted FEV1
Groups:
- Aspirin-sensitive Asthmatics: Asthma patients with aspirin exacerbated respiratory disease
Arm/Group | Aspirin-sensitive Asthmatics
Number analyzed (Participants) | 16
change in percent predicted FEV1 | 12 (1.1)

ADVERSE EVENTS:
Time Frame: 12 hours
Description: patients will be assessed for adverse reactions during their aspirin challenge (standard of care)
Arm/Group | Aspirin-sensitive Asthmatics | Aspirin-tolerant Asthmatics
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/13
Other Adverse Events (participants affected / at risk) | 0/16 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes